CLINICAL TRIAL: NCT00054405
Title: A Phase I Investigation of IL-12 (NSC 672423)/Pulse IL-2 (Aldesleukin) in Children With Persistent and/or Refractory Neuroblastoma (13623)
Brief Title: Interleukin-12 and Interleukin-2 in Treating Patients With Refractory or Recurrent Neuroblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00024; NANT 2001-01; CDR0000270447; P01CA081403 (NIH); CDR0000270447 (Registry Identifier: PDQ (Physician Data Query)); NCT00065494 (obsolete NCT alias)
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Recurrent Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Interleukin-12 Subunit p35; Interleukin-12; aldesleukin; Interleukin-2

ARMS (1):
- Treatment (IL-12, aldesleukin) (Experimental): Cohort A: Patients receive interleukin-12 (IL-12) IV over 5-15 seconds on days 1, 3, 5, 8, 10, and 12.
  Cohort B: Patients receive interleukin-2 (IL-2) IV over 15 minutes twice daily on days 1 and 8 and IL-12 IV as in cohort A.
  Treatment in both cohorts repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Some patients may receive additional courses at the discretion of the principal investigator.
  Cohorts of 3-6 patients in both cohorts receive escalating doses of IL-2 and IL-12 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  Once the MTD is determined, an additional cohort of 8 patients receives IL-12 and IL-2 at the MTD.
  Interventions: Biological: recombinant interleukin-12; Biological: aldesleukin

INTERVENTIONS:
Biological: recombinant interleukin-12 — Given IV
  Other Names: cytotoxic lymphocyte maturation factor; IL-12; interleukin-12; natural killer cell stimulatory factor; Ro 24-7472
Biological: aldesleukin — Given IV
  Other Names: IL-2; Proleukin; recombinant human interleukin-2; recombinant interleukin-2

SUMMARY:
Phase I trial to compare the effectiveness of interleukin-12 with or without interleukin-2 in treating young patients who have refractory or recurrent neuroblastoma. Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing. Combining interleukin-2 with interleukin-12 may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Define the maximum tolerated dose and dose-limiting toxicity of interleukin-12 with or without interleukin-2 in patients with refractory or recurrent neuroblastoma.

II. Determine, preliminarily, the antitumor effect of interleukin-12 with or without interleukin-2 in these patients.

III. Evaluate the immunoregulatory activity of interleukin-12 with or without interleukin-2 in these patients.

IV. Evaluate the antiangiogenic activity of interleukin-12 with or without interleukin-2 in these patients.

OUTLINE: This is a dose-escalation, multicenter study. Patients are assigned to 1 of 2 treatment cohorts.

COHORT A: Patients receive interleukin-12 (IL-12) IV over 5-15 seconds on days 1, 3, 5, 8, 10, and 12.

COHORT B: Patients receive interleukin-2 (IL-2) IV over 15 minutes twice daily on days 1 and 8 and IL-12 IV as in cohort A.

Treatment in both cohorts repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Some patients may receive additional courses at the discretion of the principal investigator.

Cohorts of 3-6 patients in both cohorts receive escalating doses of IL-2 and IL-12 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Once the MTD is determined, an additional cohort of 8 patients receives IL-12 and IL-2 at the MTD.

Patients are followed at 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of neuroblastoma

  * Histologically confirmed disease AND/OR disease defined by tumor cells in the bone marrow and elevated urinary catecholamine metabolites
* Persistent and/or refractory disease, with at least 1 of the following:

  * Biopsy-proven residual disease at least 12 weeks after myeloablative therapy
  * Progressive disease after nonmyeloablative or myeloablative therapy
* Recurrent disease, evidenced by any of the following:

  * Biopsy-proven recurrent soft tissue disease
  * Metaiodobenzylguanidine (MIBG)-positive lesions visible on any other imaging modality or repeat MIBG obtained 2-4 weeks or more apart
  * Histologically confirmed bone marrow disease
  * Progressive or stable disease after at least 1 prior standard salvage regime
* No clinically significant pleural effusion
* ECOG 0-1
* Life expectancy >= 12 weeks
* Hepatitis A antibody negative
* Hepatitis B surface antigen negative

  * Positive hepatitis B titer allowed if patient has been immunized and has no history of disease
* Hepatitis C virus negative
* No history of congenital or acquired coagulation disorder
* Cardiac function normal by ECG
* No dyspnea at rest
* No exercise intolerance
* Oxygen saturation at least 94% by pulse oximetry
* DLCO greater than 60% of predicted
* FEV1 greater than 70% of predicted
* Negative pregnancy test
* Skull-based bony lesions without space-occupying intracranial extension are allowed
* No prior or concurrent intracranial metastatic disease to the brain parenchyma
* Not pregnant or nursing
* Fertile patients must use effective barrier contraception during and for at least 2 months after study
* No prior hematologic malignancy (including leukemia or lymphoma)
* No history of malignant hyperthermia
* No prior or concurrent autoimmune disease
* No positive direct Coombs testing
* No history of ongoing or intermittent bowel obstruction
* No active infection or other significant systemic illness
* More than 2 weeks since prior fenretinide
* More than 2 weeks since prior 13-cis-retinoic acid
* More than 2 weeks since prior filgrastim (G-CSF) or sargramostim (GM-CSF)
* More than 2 weeks since prior interferons or interleukins
* More than 2 weeks since prior cytokine-fusion proteins
* More than 2 weeks since prior IV immunoglobulin (IVIG)
* No prior interleukin-12
* No concurrent cytokines
* No concurrent fenretinide
* No concurrent 13-cis-retinoic acid
* No other concurrent immunomodulators, including:

  * G-CSF and GM-CSF
  * Interferons
  * Other interleukins
  * IVIG
* More than 4 weeks since prior chemotherapy
* No other unstable medical condition or critical illness that would preclude study participation
* More than 12 weeks since prior myeloablative chemotherapy followed by autologous stem cell transplantation:

No prior myeloablative chemotherapy followed by allogeneic bone marrow transplantation

* More than 2 weeks since prior growth hormones
* More than 4 weeks since prior systemic corticosteroids
* More than 2 weeks since prior non-corticosteroid hormonal therapy (including oral birth control pills)
* No concurrent hormonal therapy (including oral birth control pills)
* No concurrent growth hormones
* No concurrent systemic corticosteroids, except for use in life-threatening complications
* More than 4 weeks since prior radiotherapy
* No prior solid organ transplantation
* More than 4 weeks since prior investigational agents
* No other concurrent investigational agents
* No prior enrollment on COG-A3973, unless disease has progressed
* No history of hemolytic anemia
* Absolute neutrophil count at least 1,500/mm^3 [Note: Independent of growth factor or transfusion support]
* Platelet count at least 75,000/mm^3 [Note: Independent of growth factor or transfusion support]
* AST and ALT less than 2.5 times upper limit of normal
* Bilirubin less than 2.0 mg/dL
* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min OR creatinine normal
* HIV negative
* Ejection fraction at least 50% by echocardiogram or MUGA OR Fractional shortening at least 30% by echocardiogram
* No congestive heart failure
* No uncontrolled cardiac arrhythmia

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2002-12; Primary Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) assessed by Common Toxicity Criteria (CTC) | 28 days

SECONDARY OUTCOMES:
Overall response assessed by Response Evaluation Criteria for Solid Tumors (RECIST) | Up to 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jon Wigginton, Principal Investigator — New Approaches to Neuroblastoma Treatment (NANT)
Locations (14):
- United States (14):
  - New Approaches to Neuroblastoma Treatment (NANT), Los Angeles, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California at San Francisco - Comprehensive Cancer Center, San Francisco, California
  - AFLAC Cancer Center and Blood Disorders Service, Atlanta, Georgia
  - Childrens Memorial Hospital, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Michigan University Hospital, Ann Arbor, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin